CLINICAL TRIAL: NCT03408496
Title: Myofascial Release of the Trunk Physiological Chains and Muscle Stretching on Pain, Quality of Life and Functional Capacity of Patients With Fibromyalgia: Randomized Controlled Clinical Trial
Brief Title: Myofascial Release of Physiological Chains and Muscle Stretching in Patients With Fibromyalgia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidade Federal de Pernambuco (Other)
Responsible Party: Principal Investigator, Nina Bretas Bittar Schulze, Principal Investigator, Universidade Federal de Pernambuco
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NSchulze
Record Dates: First submitted 2018-01-07; First posted 2018-01-24 (Actual); Last update posted 2019-03-21 (Actual); Status verified 2018-09

CONDITIONS: Fibromyalgia
Keywords: Myofascial release; Pain; Manual therapy; Muscle stretching; Quality of life
MeSH Terms: conditions — Fibromyalgia; Pain | interventions — Myofascial Release Therapy; Muscle Stretching Exercises

STUDY DESIGN:
Intervention Model Description: Participants will be allocated in 3 groups. The myofascial release group, muscle stretching group and control group.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Myofascial release (Experimental): Eight consecutive weekly sessions lasting 40-45 minutes of myofascial release of the trunk physiological chains. The connective tissue of the flexion chain and the posterior static chain will be released. The myofascial release will be obtained through the mechanical effect produced by the friction of the therapist's hand with a surface of the patient's body, which is performed through "traces" executed with the fingers (thumb supported or middle finger on the indicator to achieve effect local) following as addressed chains. The release will be repeated until the feeling of local relaxation of the tissue.
  Interventions: Other: Myofascial release
- Muscle Stretching (Experimental): The muscle stretching protocol described by Bressan (2008) will be followed, which consists of 8 consecutive weekly sessions, lasting 40-45 minutes. In dorsal decubitus or sitting, the triceps surae, hamstring, gluteal, paravertebral, latissimocondyloideus, pectoral, trapezius and respiratory muscles will be stretched. The exercises will be performed in a series of five repetitions for 30 seconds.
  Interventions: Other: Muscle stretching
- Control (Active Comparator): It will perform only the treatment prescribed by the responsable doctor, wich can be the use of drug and/or psychological treatment, and will be followed clinically by a rheumatologist during four medical appointments to monitor medication and follow in the analgesic's diary, according the standard procedure of attending the hospital where the patients will be recruited.
  Interventions: Other: Control

INTERVENTIONS:
Other: Myofascial release — Manual therapy
  Arms: Myofascial release
Other: Muscle stretching — Muscle stretching
  Arms: Muscle Stretching
Other: Control — Medical appointment
  Arms: Control

SUMMARY:
Muscle stretching is a therapeutic technique commonly used by physiotherapists, but for the treatment of fibromyalgia it still has weak evidence to support its real effect. On the other hand, myofascial mobilization in the location of tender points, as it is the solution for the population, demonstrating effects on the improvement of the symptoms, but not yet achieving the minimal clinically important change. In this context, myofascial release guided by physiological chains, so far not studied, is presented as an alternative to improve pain and quality of life in patients with fibromyalgia because it acts in a global way and, probably, more effective.

This study evaluates the effect of myofascial release of the trunk physiological chains and muscle stretching on pain, quality of life and functional capacity of patients with fibromyalgia when compared to the control group.

ELIGIBILITY:
Inclusion Criteria:

* Confirmation of the diagnosis by rheumatologists according to the diagnostic criteria established by the American College of Rheumatology of 1990 and 2010.
* Moderate to severe pain according to the Fibromyalgia Impact Questionnaire (≥ 4).
* Prescribed treatment (drug and/or psychological) stable in the last month before the selection for those who perform.
* Patients who live in the metropolitan area of Recife - Pernambuco, Brazil.

Exclusion Criteria:

* Nonpharmacologic therapies, except for psychological treatment if prescribed by the doctor at the same time of the study.
* Skin diseases.
* Patients classified as "very active" by the International Physical Activity Questionnaire.
* Women who use intrauterine devices (IUD).
* Pregnant women.
* Patients with other associated rheumatic disease or with modified posture due to congenital anatomic alteration.
* Severe decompensated comorbidities (cancer, thyroid disease and diabetes).
* Infection, fever, hypotension, respiratory alterations limiting treatment.
* Cardiovascular event in the previous year.
* Presence of cardiac, renal or hepatic insufficiency.
* Arterial or peripheral venous insufficiency.
* Presence of a hypertrophic scar on the trunk.
* Obesity grade 3.
* Illiteracy.
* Severe psychiatric illness.

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 38 (Actual)
Dates: Start 2018-01-23 (Actual); Primary Completion 2019-02-16 (Actual); Study Completion 2019-03-19 (Actual)

PRIMARY OUTCOMES:
Pain intensity level change | Baseline, after 4 weeks since the beginning of the treatment, after 8 weeks since the beginning of the treatment, follow-up (after 12 weeks since the beginning of the treatment)
  Self reported pain intensity measured by the Visual Analog Scale, wich ranges from 0 to 10, where 0 means absence of pain and 10 means the worst pain already felt
Quality of life score change | Baseline, after 4 weeks since the beginning of the treatment, after 8 weeks since the beginning of the treatment, follow-up (after 12 weeks since the beginning of the treatment)
  Evaluated by the Fibromyalgia Impact Questionnaire, wich evaluates aspects of functional capacity, work status, psychological disturbances and physical symptoms. The total score ranges from 0 to 100, where higher scores have a worst impact of fibromyalgia on quality of life and functional capacity.

SECONDARY OUTCOMES:
Amount of analgesic ingested | Up to 12 weeks
  Measured by the analgesic diary, wich is filled weekly

CONTACTS AND LOCATIONS:
Locations (1):
- Universidade Federal de Pernambuco, Recife, Pernambuco, Brazil